CLINICAL TRIAL: NCT04751877
Title: Multicenter Open Label Phase 3 Study of Isatuximab Plus Lenalidomide and Dexamethasone With/Without Bortezomib in the Treatment of Newly Diagnosed Non Frail Transplant Ineligible Multiple Myeloma Elderly Patients (≥ 65; < 80 Years).
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Collaborators: Intergroupe Francophone du Myelome (Network); Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BENEFIT - IFM2020-05
Record Dates: First submitted 2021-02-04; First posted 2021-02-12 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Multiple Myeloma; Myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — isatuximab; Lenalidomide; Bortezomib; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Isatuximab/Lenalidomide/Dexamethasone/Bortezomib (Experimental)
  Interventions: Drug: Isatuximab; Drug: Lenalidomide; Drug: Bortezomib; Drug: Dexamethasone
- Isatuximab/Lenalidomide/Dexamethasone (Active Comparator)
  Interventions: Drug: Isatuximab; Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Isatuximab — Isatuximab by IV route, per 28 days cycle - Cycle1: 10 mg/kg on days 1, 8, 15, and 22. Cycles 2 to 12: 10 mg/kg on days 1 and 15. From cycle 13: 10 mg/kg on day 1.
Drug: Lenalidomide — Lenalidomide by oral route, per 28 days cycle - 25 mg daily on days 1-21.
Drug: Bortezomib — Bortezomib sub-cutaneous, per 28 days cycle - Cycles 1 to 12: 1.3 mg/m2 on days 1, 8, 15. Cycles 13-18: 1.3 mg/m2 on days 1, 15.
  Arms: Isatuximab/Lenalidomide/Dexamethasone/Bortezomib
Drug: Dexamethasone — Dexamethasone by oral route, per 28 days cycle - 20 mg daily on days 1, 8, 15 and 22.

SUMMARY:
Overall the issue of patients above 65-70 years of age being that it is impossible for most of them to undergo an intensive treatment like autologous stem cell transplant with little prospect of debulking effectively the bone marrow with chemotherapy, and also few possibilities to harass the bone microenvironment in the tumoral niche.

If, advanced age in frail patients is predictive of an increased risk of treatment-related toxicity, there is a growing number of elderly patients in regards to transplantation, but still fit if one considers the objectives of life characterized with prolonged survival. These patients might have the same treatment as to the transplant eligible, but without the transplant procedure. The development of immunotherapy has transformed the treatment landscape of cancer, particularly in MM, increasing the treatment possibilities with possibly fewer adverse events.

The therapeutic strategy and treatment options for NTE patients moved from melphalan-based induction regimens to lenalidomide-based associations, which is now the backbone of most treatment for NTE patients. Even though the latest melphalan, bortezomib and prednisone (MPV) association was considered somewhat effective it was not so well tolerated. Furthermore, MPV hardly prolonged PFS beyond 2 years. It was recently improved with the addition of Daratumumab, first in class anti CD38 Mab in the phase III ALCYONE.

The association lenalidomide and dexamethasone (Rd) has significantly improved the easiness of treating the NTE population and all drugs seem to be possible to combine to Rd. In that extent, proteasome inhibitors have always been one of the most impactful family of agents in MM, and as expected Bortezomib plus Rd has become a very relevant and commonly used regimen in NTE NDMM. These groundbreaking results have favored the development of 2 randomized phase 3 studies for registration of combination of antiCD38Mab (Daratumumab (Cepheus, NCT03652064), Isatuximab (Imroz, NCT03319667) +Rd +Velcade in comparison to VRd. Both studies have used as a comparator the VRd regimen which is today one of the safest, active and popular triplet based Rd regimen, approved, and therefore the best control arm possibly for these studies.

However, as much as there has been no direct head to head comparison of VRd to Dara Rd, when looking at the data from Maia it is anticipated that DRd will become a standard of care, and might challenge strongly VRd. Yet, multiple questions remain still, anticipating the change in backbone from VRd to antiCD38 +Rd becoming the new standard of care for NTE NDMM patients. The investigators have therefore planned to answer the critical question of the role of proteasome inhibitors in NTE non frail NDMM when considering anti CD38 +Rd as the backbone.

ELIGIBILITY:
Inclusion Criteria:

Must be able to understand and voluntarily sign an informed consent form

* Life expectancy > 6 months
* Subject, male or female, must be at least ≥ 65 years of age and < 80 years of age
* Must have a Newly diagnosed Multiple Myeloma requiring therapy (SLiM CRAB criteria)
* Must have measurable disease
* Must be Non Transplant Eligible Non Frail

  * Newly diagnosed and not considered candidate for high-dose hemotherapy with SCT.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1, or 2
* Adequate bone marrow function, documented within 72 hours and without transfusion 72 hours prior to the first intake of investigational product (C1J1) with no growth factor support (one week),
* Adequate organ function defined as:
* Subjects affiliated with an appropriate social security system.
* A man who is sexually active with a pregnant woman or a woman of childbearing potential must agree to use a barrier method of birth control e.g., condom with spermicidal foam/gel/film/cream/suppository during the study and for at least 5 months after the last dose of treatment, even he has had a vasectomy.
* A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

Not a female of childbearing potential Or A FCBP who must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 10 - 14 days prior to and again within 24 hours prior to starting study medication and before each cycle of study treatment.

A FCBP must understand and agree to continue abstinence from heterosexual intercourse or to use 2 reliable effective methods of contraception (a very effective method and an effective additional method) simultaneously without interruption

* All patients must understand and accept to comply with the conditions of the lenalidomide pregnancy prevention plan

Exclusion Criteria:

* Subject has a diagnosis of primary amyloidosis, monoclonal gammopathy of undetermined significance, or smoldering multiple myeloma. Monoclonal gammopathy of undetermined significance is defined by presence of serum M-protein <3 g/dL; absence of lytic bone lesions, anemia, hypercalcemia, and renal insufficiency related to the M-protein; and (if determined) proportion of plasma cells in the bone marrow of 10% or less (Kyle 2003). Smoldering multiple myeloma is defined as asymptomatic multiple myeloma with absence of related organ or tissue impairment end organ damage (Kyle 2003, Kyle 2007).
* Subject has a diagnosis of Waldenström's disease, or other conditions in which IgM M-protein is present in the absence of a clonal plasma cell infiltration with lytic bone lesions.
* Subject has prior or current systemic therapy or SCT for multiple myeloma, with the exception of an emergency use of a short course (equivalent of dexamethasone 40 mg/day for a maximum 4 days) of corticosteroids before treatment.
* Subject has a history of malignancy (other than multiple myeloma) within 3 years before the date of randomization (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or malignancy that in the opinion of the investigator, with concurrence with the Coordinator Investigator, is considered cured with minimal risk of recurrence within 3 years).
* Subject has had radiation therapy within 7 days of randomization.
* Subject has had plasmapheresis within 7 days of randomization.
* Subject is exhibiting clinical signs of meningeal involvement of multiple myeloma.
* Subject known to be seropositive for history of human immunodeficiency virus (HIV) or to have hepatitis A active infection.
* Known to have hepatitis B active or uncontrolled infection (positive HBsAg and/or HBV DNA)

  * Patient can be eligible if anti-HBc IgG positive (with or without positive anti-HBs) but HBsAg and HBV DNA are negative.

If anti-HBV therapy in relation with prior infection was started before initiation of IMP, the anti-HBV therapy and monitoring should continue throughout the study treatment period.

o • Patients with negative HBsAg and positive HBV DNA observed during screening period will be evaluated by a specialist for start of anti-viral treatment: study treatment could be proposed if HBV DNA becomes negative and all the other study criteria are still met.

• Known to have hepatitis C active infection (positive HCV RNA and negative anti-HCV) Patients with antiviral therapy for HCV started before initiation of IMP and positive HCV antibodies are eligible. The antiviral therapy for HCV should continue throughout the treatment period until seroconversion.

Patients with positive anti-HCV and undetectable HCV RNA without antiviral therapy for HCV are eligible.

* Subject has any clinically significant medical or psychiatric condition or disease (e.g., uncontrolled diabetes, acute diffuse infiltrative pulmonary disease) in the investigator's opinion, would expose the patient to excessive risk or may interfere with compliance or interpretation of the study results.
* Subject has active systemic infection and severe infections requiring treatment with a parenteral administration of antibiotics.
* Subject has clinically significant cardiac disease,
* Subject has known allergies, hypersensitivity, or intolerance to steroids, mannitol, pregelatinized starch, sodium stearyl fumarate, histidine (as base and hydrochloride salt), arginine hydrochloride, poloxamer 188, sucrose or any of the other components of study intervention that are not amenable to premedication with steroids and H2 blockers or would prohibit further treatment with these agents, monoclonal antibodies or human proteins, or their excipients.
* Known hypersensitivity, allergy to one of the study product (isatuximab, lenalidomide, bortezomib), dexamethasone or to one of the excipients
* Acute diffuse infiltrative pneumopathy, pericardial disease
* Subject has plasma cell leukemia.
* Subject has had major surgery within 2 weeks before randomization or has not fully recovered from surgery, Kyphoplasty or vertebroplasty is not considered major surgery.
* Subject has received an investigational drug (including investigational vaccines) within 14 days or 5 half-lives of the investigational drug prior to initiation of study intervention, whichever is longer, or used an invasive investigational medical device within 4 weeks before randomization or is currently enrolled in an interventional investigational study.

In case of very aggressive disease (i.e acute leukemia) delay could be shortened after agreement between sponsor and investigator, in absence of residual toxicities from previous therapy.

* Refusal to consent or protected by legal regime (under judicial protection, guardianship, trusteeship)
* Subject has contraindications to required prophylaxis for deep vein thrombosis and pulmonary embolism
* Incidence of gastrointestinal disease that may significantly alter the absorption of oral drugs.

Ages: 65 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 270 (Actual)
Dates: Start 2021-07-17 (Actual); Primary Completion 2024-06-18 (Actual); Study Completion 2027-08-17 (Estimated)

PRIMARY OUTCOMES:
Minimal Residual Disease (MRD) rate at 10-5 at 18 months | at 18 months
  Proportion of patients with a reduction tumoral mass ≥50 percent who experience a Minimal Residual Disease (MRD) 10-5 per IMWG (International Myeloma Working Group) criteria.

SECONDARY OUTCOMES:
Safety of trial treatments | Up to 5 years
  List of AE frequency (AE assessed by Common Terminology Criteria for Adverse Events (CTCAE) criteria, version 5.0)
To determine the best response to the treatment | Up to 5 years
  Per International Myeloma Working Group (IMWG) criteria
Progression Free survival | Up to 5 years
  Time to relapse or death, whatever occurs first
To determine the time to reach MRD negative rate at 10-5 | Up to 5 years
  The time from randomization to the date of the first MRD negative rate at 10-5
To determine the time to loss of MRD negative rate at 10-5 | Up to 5 years
  Time from randomization or from the date of MRD negative at 10-5 to the date of MRD positive at 10-5
To evaluate the MRD rate at 10-5 at 12 months, and yearly (and at 10-6) | Up to 5 years
  Proportion of patients with a reduction tumoral mass ≥75 percent or who has reached at least SD and with MRD negative at the previous MRD assessment who experience a Minimal Residual Disease (MRD) 10-5 per IMWG (International Myeloma Working Group) criteria.
To determine the rate of loss of MRD at 10-5 at each time point | Up to 5 years
  Proportion of patients with MRD negative at 10-5 who lose the MRD negative status at the next evaluation.
To determine the sustained MRD rate at 10-5 (similar time points) | Up to 5 years
  Proportion of patients with sustained MRD in bone marrow aspirate (< 10-5) between 2 evaluations as determined in the protocol.

CONTACTS AND LOCATIONS:
Overall Officials: LELEU Xavier, Prof., Principal Investigator — Poitiers University Hospital
Locations (1):
- CHU Poitiers, Poitiers, France

REFERENCES:
- [Derived] Leleu X, Hulin C, Lambert J, Bobin A, Perrot A, Karlin L, Roussel M, Montes L, Cherel B, Chalopin T, Slama B, Chretien ML, Laribi K, Dingremont C, Roul C, Mariette C, Rigaudeau S, Calmettes C, Dib M, Tiab M, Vincent L, Delaunay J, Santagostino A, Macro M, Bourgeois E, Orsini-Piocelle F, Gay J, Bareau B, Bigot N, Vergez F, Lebreton P, Tabrizi R, Waultier-Rascalou A, Frenzel L, Le Calloch R, Chalayer E, Braun T, Lachenal F, Corm S, Kennel C, Belkhir R, Blade JS, Joly B, Richez-Olivier V, Gardeney H, Demarquette H, Robu-Cretu D, Garderet L, Newinger-Porte M, Kasmi A, Royer B, Decaux O, Arnulf B, Belhadj K, Touzeau C, Mohty M, Manier S, Moreau P, Avet-Loiseau H, Corre J, Facon T. Isatuximab, lenalidomide, dexamethasone and bortezomib in transplant-ineligible multiple myeloma: the randomized phase 3 BENEFIT trial. Nat Med. 2024 Aug;30(8):2235-2241. doi: 10.1038/s41591-024-03050-2. Epub 2024 Jun 3. PMID 38830994